CLINICAL TRIAL: NCT02114593
Title: Evaluation of a Parent Support Program to Promote Somali Parent's and Children's Mental Health
Brief Title: Ladnaan - an Evaluation of a Parent Support Program for Somali Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Dalarna University (Other)
Responsible Party: Principal Investigator, Marie Klingberg-Allvin, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ladnaan123; Dnr 2014/048 (Other: Regional ethical board in Uppsala)
Record Dates: First submitted 2014-04-12; First posted 2014-04-15 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Mental Illness
Keywords: Mental Health; Children; Parent support program; Somali families; Sweden
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent support program (Experimental): Parent support program
  Interventions: Behavioral: Parent support program
- Standard activities (No Intervention): Standard activities

INTERVENTIONS:
Behavioral: Parent support program — Parent support program
  Arms: Parent support program

SUMMARY:
The aim of this project is to evaluate the effectiveness of a culturally adapted parenting support program for Somali parents living in Sweden on children's and parent´s mental health. In recent years the Somali population in Sweden has increased and is currently one of the largest groups among ethnic minorities. Most of the Somali people have arrived as refugees and have experienced war, trauma and conflict. Research shows that migration to a new social context/society is challenging for a family and may together with previous experiences of war, separation, create stress and mental illness. This leads to consequences such as family violence, child abuse, relational problems, drug problems and school problems for children. There is a vast knowledge on the association between parents' mental health, positive parent-child relationship and children's health and well-being. Previous studies have shown that parenting programs aimed to support parent-child relationship and/or improve parental skills have positive effects on parental mental health and on children's behavior. Most municipalities in Sweden offer their residents a structured parenting program, but these programs do not reach those of ethnic minorities. Studies show that parenting programs mainly target parents who can speak Swedish fluently and that the parenting programs are not yet culturally adapted.

DETAILED DESCRIPTION:
In recent years the Somali population in Sweden has increased and is currently one of the largest groups among ethnic minorities in Sweden (http://www.scb.se). Most of the Somali people living in Sweden have arrived as refugees and they have experienced war, trauma and conflict. Research shows that migration to a new social context/society is challenging for a family and may together with previous experiences of war, separation, create mental ill-health (Bhugra, 2004; FoU, 2008). According to several studies, refugee families have poorer health and low social status compared to the native Swedish (Bhugra, 2004). Previous studies reported that both parents and children who have experienced war and conflict suffer from stress and are at risk for mental ill-health. This stress leads to various consequences such as family violence, child abuse, relational problems between parents and children, drug problems and school problems for children (Ajdukovic, et al., 1993; James, 1997; Schimtz, et al., 2003). Experience of war and conflict has further shown to have a negative impact on parent's ability to care for their children (Jack, 2000).

There is a vast knowledge on the association between parents' mental health, positive parent-child relationship and children's health and well-being (e.g. Bremberg, 2002). Previous studies have shown that parenting programs aimed to support parent-child relationship and/or improve parental skills have positive effects on parental mental health and on children's behavior (Lindsay et al., 2011; Bjorknes et al., 2013; Stewart-Brown et al., 2011). For example, parents who have participated in parenting programs report feeling less worried, stressed and depressed (Lindsay, et al., 2011; Marcynyszyn, et al., 2011, Phelan, et al., 2012; Stewart-Brown, et al., 2004). Hence, by supporting parents in their role as parents, improvements can be seen in both parents' and children's health and well-being.

According to the Swedish governmental national strategy, parents should be offered support and knowledge on how to strengthen their parenting role (Reports, 2008). Almost all the municipalities in Sweden offer their residents a structured parenting program. However, these parenting programs do not reach all residents in the municipalities, especially those of ethnic minorities (Fabian, et al., 2006; Fabian, et al., 2004), due to language barriers and lack of information about existing parenting programs to the ethnic minorities. Studies show that parenting programs mainly target parents who can speak Swedish fluently and that the parenting programs are not culturally adapted (Kling, et al., 2010). Other international studies emphasize that single or young parents, families with low socioeconomic status or who live in deprived areas, have low attendance and high drop out of parenting program (Byrne, et al., 2013; Stewart-Brown, et al., 2011).

Attempts have been made to culturally adapt parenting programs both in USA, Australia and in Norway. According to (Cardona et al., 2012) cultural adaptation needs to comprise aspects of language, culture and context. In a study by Bjorknes, et al. ( 2013), the cultural adaptation made included not to have mixed groups with both mothers and fathers and to deliver the parenting program with help the of "link workers" of Somali and Pakistani background. While many Somali parents in Sweden do not attend or have no information about the parenting programs that exist in their municipality, the number of participating families might increase substantially if these programs are offered in Somali and are culturally adapted to Somali families' needs.

Aim The aim of the study is to evaluate the effectiveness of a parenting support program on parents' and children's mental health.

Research questions:

1. What are the effects of the parenting support program on children's mental health?
2. What are effects of the parenting support program on parents' mental health and parents' self-efficacy?
3. What is the cost effectiveness of the intervention? Methodological approach: A randomized controlled trial will be conducted with one intervention group (i.e. provision of the Connect parenting program) and one control group (i.e. 'usual activities) consisting of Somali parents living in Borlänge Municipality. When applicable, both parents will be randomized together as one family.

Intervention: the intervention consists of Connect, an already established and scientifically evaluated parent program. The program is based on attachment theory and focuses on the needs of the child/youth and the parent from an attachment perspective. Connect is a 10 week program, which addresses nine different principles on child development, parent-child relationship and challenging interaction. Parents meet together in small groups with a maximum of eight families together with group leaders for one hour sessions each week. In relation to this, parents are offered some beverages and snacks half an hour before the session. Both parents will be invited to the parenting program participation. The intervention will be held in Somali language by group leaders of Somali background. In total eight group leaders will be recruited and receive four days of Connect training course by Connect instructors. Instructors will give also mentorship during parenting program. The program will be proceeded by two sessions (6 hours) on cultural specific challenges, which will be based on the results from the qualitative study (I).

Setting and data collection: Parents will be recruited from the Social services and Somali associations in Borlänge. Several information meetings will be held in different facilities within the social services and Somali associations. Parents who are eligible and give their consent to participate will be asked to fill in the baseline data. Baseline data will be collected before randomization. The intervention will be evaluated by a semi-structured questionnaire. Outcome measures will be collected two and six months after the program has ended in the intervention group, with similar data collection times in the control group. The questionnaires will be translated into the Somali language. They will be filled out by the same parent throughout the study. If both parents participate the intervention their data will pooled if their answer is about the same child. The questionnaires will be answered at a time and location chosen by parents/children, during whom a Somali speaking researcher/person will be present in order to support parents/children in filling out the questionnaires if problems arise (e.g. when parents are illiterate). Outcomes: Primary outcome is improved children's mental health. Secondary outcomes are, improved parents' mental health, and parents' self-efficacy. The questionnaire will include information about the socio-demographic factors and is based on validated instruments.

Sample size and analyzes: A power analysis was conducted to determine the required sample size. When comparing two independent sample means, with alpha set at 0.05, and power at 0.80, we need a total sample of 128 children (I: 64 C: 64) to detect a medium difference (d =.5). These groups will be expanded to 75 per group (a total sample of 150 children) since we expect 20% loss during the follow up. Intention-to-treat will be used. This means that analyses will include all randomized parents in the groups to which they were randomly assigned, regardless of their adherence with the entry criteria, regardless of the treatment they actually received, and regardless of subsequent withdrawal from treatment or deviation from the protocol. The specific statistical analysis used with each outcome variable will be determined by the distribution of the outcome variables. Intergroup comparison will be made between the control group and intervention group.

Significance A number of studies show that many evidence-based parenting programs improve parental skills and parental mental well-being. Parents perceived to be less stressed, depressed and that they have more confident in their parenting role after undergoing parenting program. By evaluating the effectiveness of a culturally appropriate parenting program to Somali parents living in Sweden the project is attempting to contribute to the wellbeing of both children and parents with Somali background. The result will be used to inform stakeholders and policy makers and hopefully be used in other municipalities in Sweden. Furthermore, the results will be disseminated through international conferences and publication in international open-access journals

ELIGIBILITY:
Inclusion Criteria:

* Somali born parent
* Parent with children in Sweden and in the age 11-16 years old
* Parent with self-perceived stress about parenting

Exclusion Criteria:

* parent who is already participating in a parenting program
* Parent with psychiatric disorder

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2014-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Children's mental health | 2 months
  Child Behavior Checklist, CBCL is a validated instrument for measuring emotional and behavior problems among children. This instrument will be answered by parents.

SECONDARY OUTCOMES:
Parent's mental Health | 2 months
  General Health Questionnaire GHQ12 will be used to measure parent's mental Health.
Parent's sense of competence | 2 months
  Parenting sense of competence,PSOC consists of 16 items to measure efficacy and satisfaction in parenting
Children's mental health | 6 months
  Child Behavior Checklist, CBCL is a validated instrument for measuring emotional and behavior problems among children. This instrument will be answered by Children.
Parent's mental health | 6 months
  General Health Questionnaire GHQ12 will be used to measure parent's mental Health.
Parent's sense of competence | 6 months
  Parenting sense of competence (PSOC) consists of 16 items to measure efficacy and satisfaction in parenting.
Children's mental health | 2 months
  Child Behavior Checklist, CBCL is a validated instrument for measuring emotional and behavior problems among children. This instrument will be answered by Children.
Client satisfaction | 2 months
  Client Satisfaction Questionnaire (CSQ) consists of 10 items to assess and evaluate the intervention and parents' view.
Children's mental health | 6 months
  Child Behavior Checklist, CBCL is a validated instrument for measuring emotional and behavior problem among children. The instrument will be answered by parents.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Klingberg-Allvin, Ass. Prof., Principal Investigator — Karolinska Institutet
Locations (1):
- Borlänge County, Borlänge, Dalarna County, Sweden

REFERENCES:
- [Derived] Osman F, Vixner L, Flacking R, Klingberg-Allvin M, Schon UK, Salari R. Impact of a culturally tailored parenting programme on the mental health of Somali parents and children living in Sweden: a longitudinal cohort study. BMJ Open. 2021 Aug 19;11(8):e045067. doi: 10.1136/bmjopen-2020-045067. PMID 34413097
- [Derived] Nystrand C, Sampaio F, Hoch JS, Osman F, Feldman I. The cost-effectiveness of a culturally tailored parenting program: estimating the value of multiple outcomes. Cost Eff Resour Alloc. 2021 Apr 23;19(1):23. doi: 10.1186/s12962-021-00278-4. PMID 33892740
- [Derived] Osman F, Salari R, Klingberg-Allvin M, Schon UK, Flacking R. Effects of a culturally tailored parenting support programme in Somali-born parents' mental health and sense of competence in parenting: a randomised controlled trial. BMJ Open. 2017 Dec 7;7(12):e017600. doi: 10.1136/bmjopen-2017-017600. PMID 29222136